## **COVER PAGE**

## TITLE: Analysis of Balance and Functional Hop Tests in Athletes with Lower Extremity Injuries by Dual Task Study

## NCT05484778

**Document Date: 03.06.2021** 

## 1. Statistical Plan

Statistical analysis was made with IBM SPSS 22 package program. Shapiro Wilk test was used to evaluate the fit for normal distribution. It was found that the data showed normal distribution. Repeated measures ANOVA analysis was used for group comparisons of the variables. Before-after comparisons without group separation

Paired sample T-test was used for the level of statistical significance was taken as p 0.05. In the statistical analysis, the before after comparison applied to all participants without group discrimination was used to support interpretation of the significance of the comparisons made between groups.